CLINICAL TRIAL: NCT00228098
Title: Smoking Cessation Intervention After Stroke or Transient Ischaemic Attack. A Randomised Controlled Trial
Brief Title: Smoking Cessation Intervention After Stroke or Transient Ischaemic Attack.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Odense University Hospital (Other)
Collaborators: Danish Heart Foundation (Other); Hjernesagen (Unknown); Funen County (Unknown)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: VF 20040136
Record Dates: First submitted 2005-09-26; First posted 2005-09-28 (Estimated); Last update posted 2005-09-28 (Estimated); Status verified 2005-09

CONDITIONS: Stroke; Transient Ischemic Attack
MeSH Terms: conditions — Stroke; Ischemic Attack, Transient

INTERVENTIONS:
Behavioral: Smoking cessation

SUMMARY:
Patients with stroke or transient ischemic attach should receive advise on smoking cessation. It is however unknown if an intensive smoking cessation program is better than ordinary advise on smoking cessation during hospitalisation for stroke or transient ischemic attack.

The aim of the study was to assess if an intensive smoking cessation program made more patients stop smoking after stroke or transient ischemic attack.

DETAILED DESCRIPTION:
Patients with stroke or transient ischemic attach should receive advise on smoking cessation. It is however unknown if an intensive smoking cessation program is better than ordinary advise on smoking cessation during hospitalisation for stroke or transient ischemic attack.

The aim of the study was to assess if an intensive smoking cessation program made more patients stop smoking after stroke or transient ischemic attack.

Patients with stroke or transient ischemic attack are admitted to the department of neurology at Odense University hospital. Patient who are smokers on admission and age < 76 years, inhabitants in Funen County and with symptoms developed before admission will be offered participation in the study unless they have severe stroke, stroke more than 3 weeks before admission, other severe disease or unable to participate.

Study participants will be randomised to either usual short advise on smoking cessation or an intensive smoking cessation program. All participants will be followed-up for 6 months with regard to smoking habits.

ELIGIBILITY:
Inclusion Criteria:

* Age < 76 years
* Inhabitant in Funen County
* Acute stroke or transient ischemic attack
* Symptoms with onset before admission
* Current smoker on admission

Exclusion Criteria:

* Severe stroke
* Current stroke onset more than 3 weeks before admission
* Other severe disease
* Unable to participate

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300
Dates: Start 2005-02; Study Completion 2007-02

PRIMARY OUTCOMES:
Smoking cessation rate

CONTACTS AND LOCATIONS:
Overall Officials: Søren Bak, MD, PhD, Principal Investigator — Department of Neurology, Odense University Hospital. 5000 Odense C. Denmark
Locations (1):
- Department of Neurology, Odense, Funen, Denmark